CLINICAL TRIAL: NCT06601244
Title: Pharmacokinetic Study of DALBAVANCINE in the Treatment of Biliary Complications During Liver Transplantation
Brief Title: Pharmacokinetic Study in the Biliary Complications During Liver Transplantation
Acronym: DALBATRANS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0165
Record Dates: First submitted 2024-08-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; Biliary complications; DALBAVANCINE; Pharmacokinetics
MeSH Terms: interventions — Pharmacogenomic Variants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pharmacokinetic — Biliary and blood concentration of the DALBAVANCINE

SUMMARY:
Liver transplantation is the last treatment for severe liver diseases such as advanced cirrhosis or fulminant hepatitis. This is a heavy treatment can be associated with numerous complications, particularly biliary ones.

The management of biliary complications is mixed, combining endoscopic treatment with biliary protheses and antibiotics.

A cohort study carried out at the Grenoble Alpes University Hospital showed a high prevalence of Enterococcus Faecium during these biliary complications. This epidemiology complicates the treatment, because it presents a natural resistance to cephalosporins and penicillin (60% of resistance to amoxicillin in Grenoble hospital), the first line treatment for biliary infection.

Antibiotic used to treat this infection can be DALBAVANCIN, which are compatible with outpatient follow-up.

Although the results are interesting in term of efficacy, no study has investigated the biliary diffusion of this antibiotic.

DETAILED DESCRIPTION:
This is a prospective observational descriptive monocentric study. As the biliary and blood samples taken are not part of standard patient management, this is a type 3 study involving human subjects.

In order to ascertain the value of antibiotic therapy with DALBAVANCINE for the treatment of biliary complications, it is important first to study the pharmacokinetics of these antibiotics to confirm their proper distribution at this site.

As concerns the study population, all liver transplant patients with biliary complications are eligible for inclusion. After diagnosis of a biliary complication and inclusion, the patient undergoes biliairy drainage (endoscopic or radiological) with bacteriological examination and antibiotic dosage in bile and blood.

Biliary drainage consists of placing biliary protheses repeatedly every 2 months for a year of follow-up. Endoscopic retrograde cholangiopancreatography allow an access to the biliary duct to change protheses and make bacteriological, mycological and antibiotic sample.

The antibiotic treatment consists of one perfusion of 1500 mg of DALBAVANCINE at J1, J7 and M2 after the biliary complication.

Plasma and biliary assays will be checked at M2 and M4 of treatment. These tests will be carried out at the time of changing biliary stents, which are part of routine care for these patients.

Clinical, biological and morphological trends are monitored for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Social security coverage
* Liver transplant recipient
* Hospitalized at CHUGA
* Presenting biliary complications following liver transplantation, confirmed morphologically by ultrasound, CT scan, or liver MRI:

  * Biliomas / bilioperitoneum
  * Hepatic abscess as described by the radiologist
* Undergoing biliary endoscopy or radiological drainage following the initiation of antibiotic therapy (between H0-H96 and 6 weeks +/- 2 weeks)
* Having expressed their non-opposition to participate in this study.

Exclusion Criteria:

* Patients under guardianship or deprived of liberty. Persons referred to in Articles L1121-5 to L1121-8 of the Public Health Code.
* Patients not affiliated with social security.
* Contraindication to the use of DALBAVANCIN.

Secondary exclusion criteria:

- Discontinuation of antibiotic therapy before the completion of biliary dosage measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic or biliary tract infection requiring prolonged antibiotic therapy with DALBAVANCINE.
  Patients who have liver transplantation complicated by a bilioma or liver abscess.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Description of biliary diffusion of dalbavancin | At Month 2
  Measurement of DALBAVANCIN concentration in bile at Month 2

SECONDARY OUTCOMES:
Description of the proportion of patients showing good clinical progress at Month 2 and Month 6. | at Month 2 and Month 6
  Good clinical progress is defined by the presence of 3 out of the following 3 criteria:
  * Disappearance of fever (T<38°C) or absence of fever spikes at Month 2 and Month 6 (in the absence of post-procedural biliary complications) or during follow-up.
  * Disappearance/regression of abdominal pain or absence of new abdominal pain at Month 2 and Month 6 after the endoscopic procedure (excluding post-procedural complications) or during follow-up (in the absence of another cause explaining the pain).
  * Disappearance/regression of jaundice or absence of new cutaneous-mucous jaundice at Month 2 and Month 6 after the endoscopic procedure or during follow-up (in the absence of another cause explaining the appearance of cutaneous-mucous jaundice).
Description of the proportion of patients showing good biological progress at Month 2 and Month 6. | at Month 2 and Month 6
  Good biological progress is defined by 3 out of the following 4 criteria:
  * Decrease in CRP by 50 mg/L, or a 20% decrease in CRP if the initial CRP is below 50 mg/L during follow-up at Month 2 and Month 6.
  * 50% decrease or normalization of bilirubin during follow-up at Month 2 and Month 6.
  * 50% decrease in cytolysis and cholestasis during follow-up at Month 2 and Month 6.
  * Disappearance of the causative pathogen in bile samples at 2 months after starting antibiotics.
Description of the proportion of patients showing good morphological progress at Month 2 and Month 6. | at Month 2 and Month 6
  Good morphological progress is defined by:
  - Regression of bilioma or abscess size by >50% or 2 cm at 2 months of treatment (compared to the initial imaging at the time of complication) or disappearance of bilioma or hepatic abscess at 2 or 6 months.
Record the occurrence of serious adverse events to evaluate the tolerance of the antibiotic therapy. | at Month2, Month 4 and Month 6
  Poor antibiotic tolerance is defined by the occurrence of clinical or biological side effects summarized in the product characteristics classified as frequent in the VIDAL: diarrhea, nausea, headaches, asthenia, dizziness.
Description of the antibiotic concentrations in bile relative to the MIC of the causative pathogens at Month 2. | at Month 2
  Measurement of DALBAVANCIN concentration, which must be greater than 10 times the MIC to be considered effective.
Evaluation of the biliary concentration of DALBAVANCIN in comparison with the plasma concentration. | at Month 2 and Month 4
  Calculation of the ratio between biliary and plasma concentrations of DALBAVANCIN
Evaluation of the effectiveness of DALBAVANCIN antibiotic treatment at Month 2 and Month 6. | at Month2 and Month 6
  * Description of the proportion of patients showing good clinical, morphological, and biological progress at Month 2 according to the plasma and biliary concentration ratio at Month 2, and the biliary concentration to MIC ratio of the causative pathogen at Month 2.
  * Description of the proportion of patients showing good clinical, morphological, and biological progress at Month 6 according to the plasma and biliary concentration ratio at Month 2, and the biliary concentration to MIC ratio of the causative pathogen.

CONTACTS AND LOCATIONS:
Overall Officials: Salomé GALLET, MD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- University Hospital Of Grenoble, Grenoble, France